CLINICAL TRIAL: NCT00900328
Title: A Pilot Project to Study the Expression of c-MET and p53 in Resected Lung Adenocarcinoma Specimens
Brief Title: Study of Tumor Samples From Patients With Lung Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150607; CDR0000614602 (Registry Identifier: NCI Physician Data Query); NCI-2009-00451 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; recurrent non-small cell lung cancer; stage 0 non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biomarkers in resected AC specimens): Previously collected tissue samples from patients enrolled in CALGB 140202 are assessed for mutation analysis of c-Met, EGFR, Kras, p53, and c-CBL via standard PCR and sequencing; gene amplification of c-Met via real time quantitative PCR; LOH analysis of c-CBL; expression levels of met/HGF protein in serum via ELISA; and expression levels of c-Met, EGFR, p53, c-CBL, DUB3, ALK, and EMT via IHC.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative Studies

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at tumor samples from patients with lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the correlation between c-Met expression, mutation and amplification, with stage and overall survival in patients with adenocarcinoma (AC) of the lung.

Secondary

* To determine the correlation with epithelial mesenchymal transition (EMT), EGFR mutations and expression, Kras mutations, p53 mutations, c-CBL protein expression, mutation, loss of heterozygosity (LOH), DUB3 expression & regulation, and ALK translocation, with respect to survival.
* To determine the correlation with circulating c-Met and HGF in AC and evaluate prognostic implications of circulating markers in AC of lung.
* To determine (when available) levels of circulating Met and HGF in serum before and after surgery.

OUTLINE: This is a multicenter study.

Previously collected tissue samples from patients enrolled in CALGB 140202 are assessed for mutation analysis of c-Met, EGFR, and K-ras. DNA is examined by PCR, followed by agarose gel electrophoresis; gene amplification of c-Met is examined by real time quantitative PCR; met/HF protein in serum is examined by ELISA; and c-Met, EGFR, p53, c-CBL, DUB3 enzyme, and ALK, and epithelial mesenchymal transition examined by IHC.

ELIGIBILITY:
Inclusion Criteria:

* Registration to Cancer and Leukemia Group B (CALGB) 140202
* Institutional Review Board (IRB) review and approval at the institution where the laboratory work will be performed is required
* Informed consent: the CALGB does not require that a separate consent form be signed for this study

  * The subject population to be studied in this protocol includes patients selected from CALGB 140202; all such patients have signed a written informed consent document meeting all federal, state, and institutional guidelines as part of entry into that trial
  * All samples to be studied were obtained and stored as part of CALGB 140202; the material and data obtained from the patient's protocol record will be used to obtain appropriate clinical information; in no instance will the patient be contacted directly
  * There should be no physical, psychological, social, or legal risks associated with this study; no invasive procedures are recommended or requested
  * All appropriate and necessary procedures will be utilized to maintain confidentiality; all patients who have had samples submitted for analysis will have their CALGB study number used to identify specimens
  * This study does not require direct patient contact and no specific risk or benefits to individuals involved in the trial are anticipated; it is likely, however, that the information gained will substantially help similar patients in the future

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung adenocarcinoma enrolled on CALCB 140202
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2008-09; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
c-Met expression | Baseline
  The correlation of c-Met expression and stage will be tested using Fisher's exact test. The proportions of c-Met overexpressed in stage I and stage II or higher will be estimated as well as the confidence intervals. The correlation of c-Met expression and survival will be tested using log rank test. The hazard ratio and its confidence interval will be estimated using a Cox model with a single predictor. Summary statistics will be provided for all c-Met measures.

SECONDARY OUTCOMES:
EMT expression | Baseline
  The correlation of EMT, EGFR mutations and expression, Kras mutations, p53 mutations, c-CBL protein expression, mutation, and LOH, DUB3 expression, and ALK translocation, circulating c-Met and HGF with respect to survival will be evaluated by Cox model with these markers as continuous predictors or by log rank test with these biomarkers dichotomized at certain cutoff points, such as median or ad hoc optimal cutoff points.
Mutations in EGFR, Kras, p53, and c-CBL | Baseline
  The correlation of EMT, EGFR mutations and expression, Kras mutations, p53 mutations, c-CBL protein expression, mutation, and LOH, DUB3 expression, and ALK translocation, circulating c-Met and HGF with respect to survival will be evaluated by Cox model with these markers as continuous predictors or by log rank test with these biomarkers dichotomized at certain cutoff points, such as median or ad hoc optimal cutoff points.
c-CBL expression and LOH | Baseline
  The correlation of EMT, EGFR mutations and expression, Kras mutations, p53 mutations, c-CBL protein expression, mutation, and LOH, DUB3 expression, and ALK translocation, circulating c-Met and HGF with respect to survival will be evaluated by Cox model with these markers as continuous predictors or by log rank test with these biomarkers dichotomized at certain cutoff points, such as median or ad hoc optimal cutoff points.
DUB3 expression and regulation | Baseline
  The correlation of EMT, EGFR mutations and expression, Kras mutations, p53 mutations, c-CBL protein expression, mutation, and LOH, DUB3 expression, and ALK translocation, circulating c-Met and HGF with respect to survival will be evaluated by Cox model with these markers as continuous predictors or by log rank test with these biomarkers dichotomized at certain cutoff points, such as median or ad hoc optimal cutoff points.
ALK Translocation | Baseline
  The correlation of EMT, EGFR mutations and expression, Kras mutations, p53 mutations, c-CBL protein expression, mutation, and LOH, DUB3 expression, and ALK translocation, circulating c-Met and HGF with respect to survival will be evaluated by Cox model with these markers as continuous predictors or by log rank test with these biomarkers dichotomized at certain cutoff points, such as median or ad hoc optimal cutoff points.
Circulating c-Met and HGF in AC | Baseline
  The correlation of EMT, EGFR mutations and expression, Kras mutations, p53 mutations, c-CBL protein expression, mutation, and LOH, DUB3 expression, and ALK translocation, circulating c-Met and HGF with respect to survival will be evaluated by Cox model with these markers as continuous predictors or by log rank test with these biomarkers dichotomized at certain cutoff points, such as median or ad hoc optimal cutoff points.
Prognostic implications of circulating markers in AC of lung | Baseline
Levels of circulating Met and HGF in serum before and after surgery (when available) | At time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Salgia, MD, PhD, Study Chair — University of Chicago
Locations (1):
- University of Chicago, Boston, Massachusetts, United States